CLINICAL TRIAL: NCT04988854
Title: Using Models' Facial Expressions to Enhance Healthy Eating Behaviour in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aston University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: #1688
Record Dates: First submitted 2021-07-26; First posted 2021-08-04 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-07

CONDITIONS: Eating Behavior
Keywords: Children
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Intervention Model Description: Children were randomly assigned to one of three conditions (positive, neutral or control)
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Positive Condition (Experimental): Children were exposed to a video of adult models eating a single piece of raw broccoli whilst showing a positive facial expression (positive video)
  Interventions: Behavioral: Facial expression video
- Neutral Condition (Experimental): Children were exposed to a video of adult models eating a single piece of raw broccoli whilst showing a neutral facial expression (neutral video)
  Interventions: Behavioral: Facial expression video
- No-Food Control Condition (Experimental): Children were exposed to a video of adult models putting pens away whilst showing a neutral facial expression (no-food control video)
  Interventions: Behavioral: Facial expression video

INTERVENTIONS:
Behavioral: Facial expression video — Children are randomly allocated to one of three conditions: positive, neutral or no-food control, where they will watch either a positive, neutral, or no-food control video.

SUMMARY:
This study examined the effect of adults' facial expressions (FEs) whilst eating raw broccoli on children's acceptance and intake of a typically less preferred vegetable. Investigating others' FEs in isolation (e.g., without statements about food tastiness) will improve understanding of the role of FEs in modelling of eating and contribute to developing strategies to help children learn pleasure from nutritious foods. Based on previous literature, it was hypothesised that children's acceptance (willingness to try, and frequency of taste exposures) and intake of raw broccoli would be higher after exposure to models eating raw broccoli with positive FEs, compared to models consuming raw broccoli with neutral FEs, or a non-food control video.

DETAILED DESCRIPTION:
Research has shown that seeing positive facial expressions towards food are effective for increasing children's desire to eat foods rated as disliked. However, the effect of adults' positive facial expressions whilst eating a raw vegetable on children's acceptance and consumption of nutritious foods that are less preferred (e.g., vegetables) remains to be established. This study examined the effect of unfamiliar adult models' facial expressions eating raw broccoli on children's acceptance and consumption of raw broccoli. Children aged 4-6-year-olds were randomised to watch a video of unfamiliar adult models eating raw broccoli with a positive or neutral facial expression, or a non-food control video. Children's acceptance (willingness to try and frequency of taste exposures) and consumption of raw broccoli was assessed. Data about parent and child characteristics was provided by parents.

ELIGIBILITY:
Inclusion Criteria:

* Child must be aged 4-6-years old. Parent and child must be living in the UK.

Exclusion Criteria:

* Children with food allergies, food intolerances, or medical conditions that affect eating behaviour were not eligible to take part.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 117 (Actual)
Dates: Start 2020-10-26 (Actual); Primary Completion 2021-02-25 (Actual); Study Completion 2021-02-25 (Actual)

PRIMARY OUTCOMES:
Raw broccoli intake | 5 minutes
  Children's intake of raw broccoli (amount of grams consumed)
Willingness to try raw broccoli | 5 minutes
  Children's willingness to try raw broccoli
Frequency of taste exposures to raw broccoli | 5 minutes
  Children's number of oral taste exposures to raw broccoli

CONTACTS AND LOCATIONS:
Overall Officials: Katie Edwards, BSc, Principal Investigator — Aston University
Locations (1):
- Aston University, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Non-identifiable data will be available upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD will be available upon request.
Access Criteria: IPD will be provided when requested by researchers. The investigators will review requests.